CLINICAL TRIAL: NCT06792448
Title: Biomarkers and Outcome Predictors of Pediatric Nephrotic Syndrome: A Genetic, Transcriptomic, and Secretome Multiomics Study
Acronym: PRECISE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Fondazione La Nuova Speranza ONLUS (Unknown); ASSOCIAZIONE SINDROME NEFROSICA ITALIA (Unknown); Nephie e.V. (Unknown); NephCEurope (Unknown); European Joint Programme on Rare Diseases (EJP RD JTC 2023) (Unknown); ERKNet (Unknown)
Responsible Party: Sponsor
Other Study IDs: 5244_11.09.2024_P; EJPRD23-108 (Other Grant/Funding Number: European Joint Programme on Rare Disease (EJP RD))
Record Dates: First submitted 2024-12-11; First posted 2025-01-24 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-11

CONDITIONS: Nephrotic Syndrome Steroid-Dependent; Nephrotic Syndrome Steroid-Resistant; Nephrotic Syndrome in Children; Glomerulonephritis; Proteinuria; Hypoalbuminemia; Kidney Diseases; Chronic Kidney Disease
Keywords: Pediatric nephrotic syndrome; Idiopathic nephrotic syndrome; Steroid-resistant nephrotic syndrome; Steroid-sensitive nephrotic syndrome; Biomarkers discovery; Genetic risk factors; Epigenetic analysis; Adaptive immune system profiling; Liquid biopsy; Serum and urine proteomics; Multiomics approach; Personalized treatment; Disease progression prediction; Molecular characterization; Pediatric kidney disease
MeSH Terms: conditions — Nephrotic Syndrome; Glomerulonephritis; Proteinuria; Hypoalbuminemia; Kidney Diseases; Renal Insufficiency, Chronic; Nephrosis, Lipoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — 1. Blood samples:
     Collected for genetic analysis. Used for peripheral blood mononuclear cells (PBMC) extraction.
  2. Urine samples:
     Collected for molecular analysis. Used to evaluate protein/creatinine ratios and perform urinalysis.
  3. Serum samples:
  Collected for molecular analysis.
  These samples are collected at various stages according to the study's protocol, including onset, relapse, and remission, for use in multiomic analyses to identify molecular predictors of disease progression and treatment response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment-Naive Idiopathic Nephrotic Syndrome (INS) Patients: This cohort comprises 110 children diagnosed with idiopathic nephrotic syndrome (INS) who are treatment-naive at enrollment. The participants will receive a standard induction therapy with prednisone or prednisolone and will be followed for 12 months. During this period, blood and urine samples will be collected at various points (enrollment, 6 weeks, 6 months, and 12 months) and in cases of relapse. The goal is to monitor disease progression and classify patients based on their response to therapy, specifically identifying subtypes such as steroid-resistant, steroid-dependent, and infrequent relapsing nephrotic syndrome .
- Healthy Pediatric Control Group: This cohort consists of 40 age-matched children without nephrotic syndrome, selected from individuals undergoing minor urological surgical procedures. These participants will provide baseline control samples (blood and urine) for comparison with the INS patients' samples. This group allows researchers to identify molecular characteristics unique to INS by contrasting them with data from healthy children .
- Prevalent Idiopathic Nephrotic Syndrome (INS) Patients: This group includes 200 INS patients who have previously received treatment and are part of the larger validation phase. This cohort will be used to confirm the biomarkers and molecular profiles identified in the main cohort. The aim is to generalize findings and ensure that identified biomarkers are consistent across a broader population. Samples will be collected during relapse and remission, aligning with the study's focus on validating predictive biomarkers of disease course and therapeutic response .

SUMMARY:
Idiopathic Nephrotic Syndrome is a rare disease of the kidneys, which typically affects children. For most affected children there is the need of a prolonged treatment with drugs reducing the activity of the immune system, also resulting in many side effects. Those patients, who do not respond to treatment, are at risk of kidney damage and of dialysis or kidney transplantation. It is currently impossible to predict the response to treatment, leading to unnecessary therapies with side effects as well as unclear prognosis in the affected children. The response of the idiopathic nephrotic syndrome to medications acting on the immune system explains its important role in the occurrence of the disease.

With this study we aim to obtain predictors of the response to treatment right at the beginning of the disease, to adapt the therapy avoiding needless side effects. This will be done evaluating the blood and urine of affected children using state of the art molecular characterisation. We will evaluate the genetic predisposition, the cell trait changes and the presence of molecules in blood and urine that may affect the interaction between the immune system and the kidneys. We expect that the findings will improve treatment of children with idiopathic nephrotic syndrome and reduce the number of children suffering from unnecessary drugs related side effects.

DETAILED DESCRIPTION:
The PRECISE study (Biomarkers and Outcome Predictors of Pediatric Nephrotic Syndrome) is an innovative, multicenter research project focused on advancing our understanding of pediatric nephrotic syndrome (NS) and improving treatment outcomes for affected children across Europe. This project, which involves multiple European institutions, centers around discovering predictive biomarkers using advanced genetic, transcriptomic, and secretome multiomics methods. Nephrotic syndrome, a complex kidney disease that primarily impacts children, can lead to significant health challenges and often necessitates prolonged treatment with immunosuppressive drugs that carry side effects.

Overview of Nephrotic Syndrome

Nephrotic syndrome is characterized by symptoms such as proteinuria (excessive protein in the urine), hypoalbuminemia (low blood albumin levels), edema (swelling), and hyperlipidemia (high blood lipids). Pediatric nephrotic syndrome, known for its unpredictable nature, is categorized as Idiopathic Nephrotic Syndrome (INS) and affects around 2-7 children per 100,000 each year. While some children respond well to steroid treatment (steroid-sensitive), a significant proportion may become steroid-resistant, risking severe kidney damage that may lead to dialysis or even kidney transplant.

Why This Study is Important

Currently, it is challenging to predict which children will respond to treatment, how their disease will progress, or which children may experience repeated relapses. The standard treatment with immunosuppressive drugs, although effective for some, can bring numerous side effects, especially with prolonged use. Therefore, one of the most pressing unmet needs in pediatric nephrology is to develop early predictive biomarkers for individualized treatment plans, ultimately reducing unnecessary drug exposure and improving long-term outcomes.

The PRECISE study is designed to fill this critical gap by identifying genetic and molecular markers that can help clinicians:

1. Predict Treatment Response - Identify children who may or may not respond to steroid therapy.
2. Anticipate Disease Progression - Understand which patients are more likely to experience relapses or progress toward kidney failure.
3. Personalize Therapy - Tailor treatments based on each patient's unique biological profile to minimize side effects and maximize effectiveness.

Objectives of the Study

The primary goal of the PRECISE study is to create a predictive model for differentiating children with Steroid-Resistant Nephrotic Syndrome (SRNS) or Steroid-Dependent Nephrotic Syndrome (SDNS) from those with Infrequent Relapsing Nephrotic Syndrome (IRNS) right at the onset of the disease. This model will integrate various data sources, including omics, genetic, and clinical information, to produce a reliable "biomarker signature" that can guide therapeutic decisions from the start.

The study has several secondary objectives, including:

1. Genetic and Epigenetic Analysis - Identifying the genetic and epigenetic factors that contribute to nephrotic syndrome's pathogenesis.
2. Immune System Profiling - Understanding how adaptive immune system alterations may influence disease onset and progression.
3. Molecular Characterization - Using advanced proteomics to identify distinct protein patterns in serum and urine that differ between disease subtypes.
4. Healthy Controls Comparison - Analyzing the molecular characteristics of healthy children to enhance the accuracy of disease-specific biomarkers.

Study Design and Methodology

The PRECISE study is an open, multicenter, observational study. It will enroll a total of 310 children diagnosed with INS and an additional control group of 40 healthy children. The study is structured as follows:

1. Discovery Phase - This phase will involve 110 treatment-naive children with INS who will be followed for 12 months. During this period, biological samples will be collected at several key points, such as at the time of diagnosis, during remission, and in case of relapse. These samples will undergo extensive molecular profiling, including genetic, proteomic, and transcriptomic analyses, which will enable the identification of key biomarkers.
2. Validation Phase - In this phase, an independent cohort of 200 INS patients (prevalent cases) will be studied to confirm the reliability of biomarkers identified in the discovery phase.

Key Elements of the Study Protocol

Inclusion Criteria for Participants

For the main study group, children must be aged between 1 and 18 years and have a clinical diagnosis of idiopathic nephrotic syndrome. They should not have undergone any previous treatment for INS and must meet specific criteria for disease markers, such as proteinuria and hypoalbuminemia. A validation cohort includes children with similar characteristics but who have already been treated, while a control group comprises healthy children with no proteinuria and minor congenital kidney conditions.

Data Collection and Sampling

At each assessment visit, clinical data will be gathered, including physical exam results, medical history, vital signs, and laboratory values. Biological samples (blood and urine) will also be collected and stored at centralized biobanking facilities, with samples being analyzed for a wide range of molecular markers. The study uses high-level biostatistics and bioinformatics to interpret the complex data, aiming to provide a multidimensional view of each participant's health profile.

Analysis and Expected Outcomes

Using advanced statistical techniques and machine learning algorithms, researchers will analyze differences in genetic, immune, and molecular markers among the different patient groups. The primary endpoint is to develop molecular signatures predictive of disease progression, which can differentiate between SRNS, SDNS, and IRNS groups. Secondary endpoints include:

* Genetic Predispositions - Assessing variants in immune- and kidney-related genes that may be associated with disease progression.
* Immune Alterations - Evaluating specific immune cell types and their behaviors, which may be linked to the risk of relapse or resistance to treatment.
* Proteomic Profiles - Identifying protein patterns in blood and urine that are unique to the disease and could be used to classify disease stages and predict outcomes.

Impact and Implications

The PRECISE study represents a major step forward in pediatric nephrology by leveraging cutting-edge scientific methods to address the pressing challenges faced by children with nephrotic syndrome. By identifying biomarkers that predict treatment response and disease progression, this study can help tailor treatments to each child's needs, reducing the risk of adverse side effects and improving overall outcomes.

Consortium and Collaborating Institutions

The project is led by the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico in Milan, Italy, under the guidance of Principal Investigator Prof. Giovanni Montini. It brings together several renowned research centers and universities across Europe, each contributing unique expertise in pediatric nephrology, genetics, and molecular biology. Key partners include Heidelberg University, University Hospital of Cologne, Medical University of Gdansk, Istanbul University, and Vilnius University, along with patient advocacy organizations such as NephCEurope and various national nephrology groups.

Through this consortium, the study integrates expertise and resources from across Europe, ensuring a robust and comprehensive approach to this challenging area of pediatric medicine.

Summary

In summary, the PRECISE study is a pioneering effort to improve the diagnosis, prognosis, and treatment of pediatric nephrotic syndrome through the identification of precise molecular biomarkers. This study not only seeks to benefit children affected by nephrotic syndrome today but also lays the groundwork for future research in rare kidney diseases. By aligning clinical care with the latest in genetic and molecular science, the PRECISE study aims to provide new hope to families affected by this chronic and often debilitating condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic nephrotic syndrome (INS) with nephrotic range proteinuria (uPr/uCr ratio > 2 mg/mg).
* Hypoalbuminemia with serum albumin < 3.0 g/dL.
* Presence of edema.
* No prior treatment for idiopathic nephrotic syndrome.
* Age between 1 and 18 years at the time of enrollment.
* igned informed consent by a parent or legal guardian.

Exclusion Criteria:

* Diagnosis of congenital or infantile nephrotic syndrome (age < 1 year).
* Diagnosis of secondary nephrotic syndrome.
* Presence of glomerulonephritis, autoimmune diseases, or vasculitis.
* Lack of signed informed consent by a parent or legal guardian.
* Previous treatment with prednisone or prednisolone for nephrotic syndrome.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study participants will be selected from a population of pediatric patients with idiopathic nephrotic syndrome (INS) who are treatment-naive and present with clinical symptoms such as proteinuria, hypoalbuminemia, and edema. These patients, aged 1 to 18 years, are typically referred to specialized nephrology clinics or tertiary care centers across Europe, where they receive initial diagnosis and follow-up care.
  The participant pool is drawn from both primary recruiting centers, which are large pediatric nephrology units with established expertise in managing nephrotic syndrome, and additional collaborating centers within the European ERKNet and ESCAPE Networks. This setting ensures a broad representation of pediatric INS cases across various European regions, enhancing the study's generalizability. Additionally, a control group of age-matched children without nephrotic syndrome is included, selected from children undergoing minor urological procedures in these clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Predictive Molecular Signature of INS Progression | Up to 1 year from enrollment after initial diagnosis.
  Identification of distinct molecular characteristics predictive of the progression of idiopathic nephrotic syndrome (INS). This includes differentiating between steroid-resistant nephrotic syndrome (SRNS), steroid-dependent nephrotic syndrome (SDNS), and infrequent relapsing nephrotic syndrome (IRNS).
  Measure Type: Analysis of genetic/epigenetic background, immune status, and vesicular proteome/transcriptomic profile.
  Goal: Develop a biomarker-based predictive model that assists in early classification of INS subtypes.

SECONDARY OUTCOMES:
Genetic and Epigenetic Risk Factors | Up to 6 months from enrollment after initial diagnosis.
  Quantification of kidney- and immune-related genetic variants associated with INS incidence and disease progression.
  Measure Type: Number of risk variants in kidney and immune-related genes, along with methylation profiles showing hypomethylated and hypermethylated regions related to immune function and progression to kidney failure .
Immune System Alterations | Up to 1 year from enrollment after initial diagnosis.
  Analysis of adaptive immune system changes in INS patients. Measure Type: Proportion and absolute numbers of B and T cell subpopulations, changes in immune cell subset genes, and phosphorylation sites in primary immune cells.
  Goal: Examine immune profiles associated with disease subtypes to better understand immunologic drivers of INS .
Proteomic Patterns in Serum and Urine | Up to 1 year from enrollment after initial diagnosis.
  Identification of unique protein profiles in serum and urine that correlate with different INS subtypes.
  Measure Type: Analysis of extracellular vesicle concentration and size in urine, surface proteome of extracellular vesicles, and serum proteome characteristics in different INS groups.
  Goal: Detect specific proteomic markers linked to disease phenotype and progression .
Molecular Profile of Healthy Control Group | At a single time point during enrollment.
  Comprehensive molecular characterization of healthy children to establish a baseline for comparison with INS patients.
  Measure Type: Similar profiling as for INS patients, focusing on genetic and proteomic markers.
  Goal: Differentiate between disease-specific and baseline molecular signatures .

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Montini, Doctor of Medicine, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico

IPD SHARING:
Plan to Share IPD: No
The PRECISE study does not plan to share Individual Participant Data (IPD). This decision prioritizes the protection of participant confidentiality and aligns with the study's ethical guidelines, ensuring that sensitive genetic, transcriptomic, and proteomic information remains secure. As such, no IPD collected throughout the trial will be made available publicly or for secondary research purposes.

DOCUMENTS (1):
  • Study Protocol (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT06792448/Prot_001.pdf